CLINICAL TRIAL: NCT06319118
Title: A Clinical Study of Dihydroergotine Mesylate Extended-release Tablets for the Treatment of Drooling in Parkinson's Disease.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JD-LK2023091-I01
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Salivation in Parkinson's Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator: placebo (Placebo Comparator): control group patients, 40 cases
  Interventions: Drug: Placebo
- Experimental: dihydroergotine mesylate sustained-release tablets (Experimental): treatment group patients, 80 cases
  Interventions: Drug: dihydroergotine mesylate sustained-release tablets

INTERVENTIONS:
Drug: Placebo — placebo + usual care, placebo 5 mg daily; 2.5mg 2 times daily, after breakfast and dinner.
  Arms: Placebo Comparator: placebo
Drug: dihydroergotine mesylate sustained-release tablets — Dihydroergotine mesylate extended-release tablets + conventional treatment, dihydroergotine mesylate sustained-release tablets 5mg daily; 2.5mg 2 times daily, after breakfast and dinner.
  Arms: Experimental: dihydroergotine mesylate sustained-release tablets

SUMMARY:
Objective: To evaluate the efficacy and safety of dihydroergotine mesylate extended-release tablets for salivation in Parkinson's disease Study content: Using a randomized, double-blind, placebo-controlled study design, 120 patients with Parkinson's disease and cognitive impairment were enrolled, and the treatment was followed up for 12 weeks: dihydroergotine mesylate sustained-release tablets + conventional treatment (treatment group patients, 80 cases), placebo + conventional treatment (control group patients, 40 cases), and the main indicators were observed: the improvement effect of dihydroergotine mesylate sustained-release tablets on PD salivation was observed, and the secondary indicators were observed: the effect of dihydroergotine mesylate sustained-release tablets on the cognitive function of PD patients was observed.

Expected results: The improvement effect of dihydroergotine mesylate sustained-release tablets on PD salivation was significantly different from that of the placebo control group. The dihydroergotine mesylate sustained-release tablet group had a significant effect on the cognitive function of PD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Parkinson's disease diagnosed by the British Parkinson's Disease Brain Bank Diagnostic Criteria can come to the hospital accompanied by family members
2. drooling score using the Parkinson's Comprehensive Rating Scale (UPDRS) Part II (Item 6) ≥3;
3. MMSE ≥ 10 points (recording the patient's education level)
4. Adults over the age of 18
5. The applicant or his/her caregiver must be able to complete the record of the salivation score
6. Patients or family members voluntarily participate and sign an informed consent form.

Exclusion Criteria:

1. Patients with non-primary Parkinson's disease
2. Known allergy to dihydroergotamine mesylate
3. Drug-induced hypersalivation, such as olanzapine, antipsychotics, clonazepam and other antiepileptic drugs, as well as direct and indirect cholinergic agonists for the treatment of Alzheimer's disease and myasthenia gravis
4. BoNT treatment for saliva within the previous 3 months
5. Patients with symptomatic bradycardia, severe orthostatic hypotension, symptomatic coronary insufficiency, severe organic cardiac damage, severe liver and kidney insufficiency: including ALT≥2.5ULN (upper limit of normal value of the executive laboratory); AST≥2.5ULN (upper limit of normal for the execution laboratory); Creatinine ≥ 1.5 ULN (upper limit of normal at the execution laboratory), active psychosis, pregnancy/pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
the objective weight of saliva in patients with Parkinson's disease changed from baseline | the objective weight of saliva in patients with Parkinson's disease changed from baseline at the 4th, 8th and 12th weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Arilliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided